CLINICAL TRIAL: NCT03099304
Title: A Randomized, Double-Blind, Dose-Ranging Study of INCB018424 Phosphate Cream in Subjects With Vitiligo
Brief Title: A Study of INCB018424 Phosphate Cream in Subjects With Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-211
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2021-12-10 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Vitiligo
Keywords: Vitiligo; depigmenting disorder; topical JAK inhibitor
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ruxolitinib cream 1.5% twice daily (BID) (Experimental): Ruxolitinib cream 1.5% BID for 52 weeks, followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension.
  Interventions: Drug: Ruxolitinib cream
- Ruxolitinib cream 1.5% once daily (QD) (Experimental): Ruxolitinib cream 1.5% QD in the morning (vehicle cream in the evening) for 52 weeks, followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension.
  Interventions: Drug: Ruxolitinib cream; Drug: Vehicle cream
- Ruxolitinib cream 0.5% QD (Experimental): Ruxolitinib cream 0.5% QD in the morning (vehicle cream in the evening) for 52 weeks, followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension.
  Interventions: Drug: Ruxolitinib cream; Drug: Vehicle cream
- Ruxolitinib cream 0.15% QD (Experimental): Ruxolitinib cream 0.15% QD in the morning (vehicle cream in the evening) for 52 weeks (opportunity for re-randomization to a higher dose at Week 24 if < 25% improvement in F-VASI score), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension.
  Interventions: Drug: Ruxolitinib cream; Drug: Vehicle cream
- Vehicle BID (Placebo Comparator): Vehicle cream BID for 24 weeks, followed by re-randomization to ruxolitinib cream 1.5% BID, 1.5% QD, or 0.5% QD for Weeks 24 to 52, followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension.
  Interventions: Drug: Ruxolitinib cream; Drug: Vehicle cream

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB018424 cream
Drug: Vehicle cream — Vehicle cream is matching in appearance to ruxolitinib cream and is to be applied in the same manner as ruxolitinib cream.
  Arms: Ruxolitinib cream 0.15% QD; Ruxolitinib cream 0.5% QD; Ruxolitinib cream 1.5% once daily (QD); Vehicle BID

SUMMARY:
The purpose of this study will be to examine the efficacy, safety, and tolerability of ruxolitinib cream in subjects with vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of vitiligo.
* Vitiligo with depigmented areas including:

  * at least 0.5% of the total body surface area (BSA) on the face (0.5% BSA is approximately equal to the area of the participant's palm [without digits]) AND
  * at least 3% of the total BSA on nonfacial areas (3% BSA is approximately equal to the area of 3 of the participant's handprints [palm plus 5 digits]).
* Participants who agree to discontinue all agents used to treat vitiligo from screening through the final follow-up visit. Over-the-counter preparations deemed acceptable by the investigator and camouflage makeups are permitted.

Exclusion Criteria:

* Conditions at baseline that would interfere with evaluation of vitiligo.
* Participants who are receiving any kind of phototherapy, including tanning beds.
* Participants with other dermatologic disease besides vitiligo whose presence or treatments could complicate the assessment of repigmentation.
* Participants who have used skin bleaching treatments for past treatment of vitiligo or other pigmented areas.
* Participants who have received any of the following treatments within the minimum specified timeframes.

  * Use of any biologic, investigational, or experimental therapy or procedure for vitiligo within 12 weeks or 5 half-lives (whichever is longer) of screening.
  * Use of laser or light-based vitiligo treatments, including tanning beds, within 8 weeks of screening.
  * Use of immunomodulating oral or systemic medications (eg, corticosteroids, methotrexate, cyclosporine) or topical treatments that may affect vitiligo (eg, corticosteroids, tacrolimus/pimecrolimus, retinoids) within 4 weeks of screening.
* Use of any prior and concomitant therapy not listed above that may interfere with the objective of the study as per discretion of the investigator, including drugs that cause photosensitivity or skin pigmentation (eg, antibiotics such as tetracyclines, antifungals) within 8 weeks of screening.
* Participants with a clinically significant abnormal thyroid-stimulating hormone or free T4 at screening.
* Participants with protocol-defined cytopenias at screening
* Participants with severely impaired liver function.
* Participants with impaired renal function.
* Participants taking potent systemic cytochrome P450 3A4 inhibitors or fluconazole within 2 weeks or 5 half-lives, whichever is longer, before the baseline visit.
* Participants who have previously received JAK inhibitor therapy, systemic or topical.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (26):
- United States (26):
  - UNIVERSITY OF ALABAMA AT BIRMINGHAM (UAB), 1802 6th Ave S, Birmingham, Alabama
  - BURKE PHARMACEUTICAL RESEARCH LLC, 3633 Central Ave, Hot Springs, Arkansas
  - NORTHWEST AR CLINICAL TRIALS CENTER, PLLC/HULL DERMATOLOGY, PA, 500 S 52nd Street, Rogers, Arkansas
  - THE VITILIGO & PIGMENTATION INSTITUE OF SOUTHERN CALIFORNIA, 5670 Wilshire Boulevard, Los Angeles, California
  - DERMATOLOGY RESEARCH ASSOCIATES- LOS ANGELES, 8930 S Sepulveda Blvd, Los Angeles, California
  - DERMATOLOGY SPECIALISTS, 3629 Vista Way, Oceanside, California
  - CLINICAL RESEARCH CENTER OF CT, 27 Hospital Avenue, Danbury, Connecticut
  - LEAVITT MEDICAL ASSOCIATES OF FLORIDA INC/ AMERIDERM RESEARCH, 725 W Granada Blvd, Ormond Beach, Florida
  - EMORY UNIVERSITY, 1525 Clifton Road, Atlanta, Georgia
  - NORTHWESTERN UNIVERSITY, 676 N Saint Clair, Chicago, Illinois
  - DAWES FRETZIN CLINICAL RESEARCH GROUP, 8103 Clearvista Parkway, Indianapolis, Indiana
  - DS RESEARCH, 2241 Green Valley Road, New Albany, Indiana
  - TULANE UNIVERSITY, 1415 Tulane Avenue, New Orleans, Louisiana
  - Tufts Medical Center, 260 Tremont Street, Boston, Massachusetts
  - UNIVERSITY OF MASSACHUESETTS, 364 Plantation Street, Worcester, Massachusetts
  - HAMZAVI DERMATOLOGY, 3031 W Grand Blvd, Detroit, Michigan
  - WASHINGTON UNIVERSITY SCHOOL OF MEDICINE DERMATOLOGY, 969 N. Mason Road, St Louis, Missouri
  - ACTIVMED PRACTICES & RESEARCH, INC, 110 Corporate Drive, Portsmouth, New Hampshire
  - ICAHN SCHOOL OF MEDICINE AT MOUNT SINAI MEDICAL CENTER- DERMATOLOGY ASSOCIATES, 5 E 98th Street, New York, New York
  - WAKE FOREST UNIVERSITY HEALTH SCIENCES, Medical Center Boulevard, Winston-Salem, North Carolina
  - CENTRAL SOONER RESEARCH, 900 N Porter Ave, Norman, Oklahoma
  - RHODE ISLAND HOSPITAL, 593 Eddy Street, Providence, Rhode Island
  - ARLINGTON RESEARCH CENTER, INC., 711 East Lamar Boulevard, Arlington, Texas
  - MENTER DERMATOLOGY RESEARCH INSTITUTE, 3900 Junius Street, Dallas, Texas
  - UNIVERSITY OF TEXAS SOUTHWESTERN MEDICAL CENTER, DEPARTMENT OF DERMATOLOGY, 5323 Harry Hines Blvd, Dallas, Texas
  - THE DERMATOLOGY AND LASER CENTER OF SAN ANTONIO, 7810 Louis Pasteur, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howell MD, Kuo FI, Rumberger B, Boarder E, Sun K, Butler K, Harris JE, Grimes P, Rosmarin D. Baseline Levels of Circulating Inflammatory Biomarkers Stratify Patients with Vitiligo Who Significantly Repigment after Treatment with Ruxolitinib Cream. JID Innov. 2023 Sep 13;3(6):100230. doi: 10.1016/j.xjidi.2023.100230. eCollection 2023 Nov. PMID 37840766
- [Derived] Rosmarin D, Pandya AG, Lebwohl M, Grimes P, Hamzavi I, Gottlieb AB, Butler K, Kuo F, Sun K, Ji T, Howell MD, Harris JE. Ruxolitinib cream for treatment of vitiligo: a randomised, controlled, phase 2 trial. Lancet. 2020 Jul 11;396(10244):110-120. doi: 10.1016/S0140-6736(20)30609-7. PMID 32653055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 157 participants with vitiligo were treated at 26 study centers in the United States.
Pre-assignment Details: 157 participants were randomized to receive 1 of 4 dose strengths of ruxolitinib cream (0.15% once daily [QD], 0.5% QD, 1.5% QD, 1.5% twice daily [BID]) or vehicle during the 24-week, double-blind (DB), vehicle-controlled treatment period. After the DB period, 11 participants remained on 0.15% QD, and 42 participants who met criteria were re-randomized to 1 of the 3 higher active blinded treatment groups. All other participants remained on the same treatment regimen through Week 52.
Groups:
- Vehicle Twice Daily (BID): Vehicle cream BID for 24 weeks (double-blind, vehicle-controlled treatment period), followed by re-randomization to ruxolitinib cream 1.5% BID, 1.5% once daily (QD), or 0.5% QD for Weeks 24 to 52 (continued double-blind treatment period), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Ruxolitinib Cream 0.15% QD: Ruxolitinib cream 0.15% QD in the morning (vehicle cream in the evening) for 24 or 52 weeks. Those who did not achieve a 25% improvement in F-VASI score were re-randomized to receive ruxolitinib cream 0.5% QD in the morning (vehicle cream in the evening), 1.5% QD in the morning (vehicle cream in the evening), or 1.5% BID for Weeks 24 to 52 (continued double-blind treatment period). All participants applied ruxolitinib cream 1.5% BID in the 104-week open-label extension period.
- Ruxolitinib Cream 0.5% QD: Ruxolitinib cream 0.5% QD in the morning (vehicle cream in the evening) for 52 weeks (combined vehicle-controlled and continued double-blind periods), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Ruxolitinib Cream 1.5% QD: Ruxolitinib cream 1.5% QD in the morning (vehicle cream in the evening) for 52 weeks (combined vehicle-controlled and continued double-blind periods), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Ruxolitinib Cream 1.5% BID: Ruxolitinib cream 1.5% BID for 52 weeks (combined vehicle-controlled and continued double-blind periods), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Cross-over: Participants who were randomized to vehicle cream BID or to ruxolitinib cream 0.15% QD in the morning (vehicle cream in the evening) on Day 1 of the double-blind, vehicle-controlled treatment period and received ruxolitinib cream 1.5% BID in the 104-week open-label extension period.
Period: DB Period: Day 1 to Week 24
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID | Cross-over
Started | 32 | 31 | 31 | 30 | 33 | 0
Completed | 27 | 26 | 30 | 26 | 30 | 0
Not Completed | 5 | 5 | 1 | 4 | 3 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Reason not specified | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0 | 2 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0 | 0
Period: DB Period: Weeks 24 to 52
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID | Cross-over
Started | 0 (Vehicle cream was not used after Week 24. After the 24-week DB period, participants who met criteria were re-randomized to 1 of the 3 higher active blinded treatment groups.) | 11 (These participants continued on the initial 0.15% QD treatment.) | 45 (Total participants included those initially randomized to 0.5% QD and those re-randomized from vehicle cream and 0.15% QD to 0.5% QD.) | 44 (Total participants included those initially randomized to 1.5% QD and those re-randomized from vehicle cream and 0.15% QD to 1.5% QD.) | 47 (Total participants included those initially randomized to 1.5% BID and those re-randomized from vehicle cream and 0.15% QD to 1.5% BID) | 0
Completed | 0 | 10 | 43 | 37 | 45 | 0
Not Completed | 0 | 1 | 2 | 7 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 1 | 0
Not completed — Reason not specified | 0 | 0 | 0 | 1 | 0 | 0
Period: 104-week Open-Label Extension Period
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID | Cross-over
Started | 0 | 0 | 28 (These participants were initially randomized to receive ruxolitinib cream 0.5% QD on Day 1 and entered the Extension Period.) | 21 (These participants were initially randomized to receive ruxolitinib cream 1.5% QD on Day 1 and entered the Extension Period.) | 28 (These participants were initially randomized to receive ruxolitinib cream 1.5% BID on Day 1 and entered the Extension Period.) | 46 (These participants were initially randomized to receive ruxolitinib cream 0.15% QD or vehicle on Day 1.)
Completed | 0 | 0 | 11 | 8 | 12 | 23
Not Completed | 0 | 0 | 17 | 13 | 16 | 23
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2 | 1 | 6
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 9 | 10 | 13 | 15
Not completed — Other Reason not specified | 0 | 0 | 4 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID | Total
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33 | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.3 (13.11) | 45.1 (11.46) | 53.8 (14.34) | 46.7 (11.73) | 49.5 (12.28) | 48.3 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 12 | 19 | 15 | 84
  Male | 12 | 13 | 19 | 11 | 18 | 73
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 10 | 6 | 6 | 6 | 5 | 33
  Not Hispanic or Latino | 21 | 22 | 23 | 21 | 27 | 114
  Not Reported | 1 | 2 | 1 | 3 | 0 | 7
  Unknown | 0 | 0 | 0 | 0 | 1 | 1
  Captured as "Other" | 0 | 1 | 1 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 26 | 29 | 25 | 23 | 29 | 132
  Black/African-American | 5 | 0 | 4 | 2 | 3 | 14
  Asian | 1 | 0 | 1 | 2 | 1 | 5
  Mexican | 0 | 1 | 0 | 0 | 0 | 1
  Nigerian/West African | 0 | 1 | 0 | 0 | 0 | 1
  Cuban | 0 | 0 | 1 | 0 | 0 | 1
  Spanish | 0 | 0 | 0 | 1 | 0 | 1
  Hispanic | 0 | 0 | 0 | 1 | 0 | 1
  Caucasian, Black, and Asian | 0 | 0 | 0 | 1 | 0 | 1
Facial Body Surface Area (F-BSA) Involvement [Mean (Standard Deviation); unit: percentage of facial surface area] — F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically and laterally from the corner of the mouth to the tragus. The area "Face" did not include the surface area of the lips, scalp, ears, or neck, but included the nose and eyelids.
  percentage of facial surface area | 1.44 (0.838) | 1.35 (0.858) | 1.40 (0.760) | 1.67 (0.953) | 1.55 (0.892) | 1.48 (0.858)
Total Body Surface Area (T-BSA) Involvement [Mean (Standard Deviation); unit: percentage of total body surface area] — T-BSA involvement was the proportion of the body surface area with vitiligo. The body was divided into the following 6 separate and mutually exclusive sites: (1) head/neck, (2) hands, (3) upper extremities (excluding hands), (4) trunk, (5) lower extremities (excluding feet), and (6) feet.
  percentage of total body surface area | 23.54 (20.960) | 17.56 (10.925) | 22.96 (21.449) | 24.81 (20.056) | 21.46 (16.820) | 22.05 (18.377)
Face Vitiligo Area Scoring Index (F-VASI) [Mean (Standard Deviation); unit: scores on a scale] — F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA; assessed by the Investigator) and the degree of depigmentation: 0% (no depigmentation), 10% (specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), 100% (no pigment). F-VASI was derived by multiplying the vitiligo involvement values by the percentage of affected skin for each facial site and summing all values (range: 0-3; lower scores indicate increased improvement).
  scores on a scale | 1.21 (0.845) | 1.19 (0.754) | 1.22 (0.705) | 1.45 (0.980) | 1.26 (0.807) | 1.26 (0.817)
Total Body Vitiligo Area Scoring Index (T-VASI) [Mean (Standard Deviation); unit: scores on a scale] — T-VASI was measured by the percentage of vitiligo involvement from all body regions (percentage of BSA; assessed by the Investigator) and the degree of depigmentation: 0% (no depigmentation), 10% (specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), 100% (no pigment). T-VASI was derived by multiplying vitiligo involvement values by the percentage of affected skin for each site and summing all values (range: 0-100; lower scores=increased improvement).
  scores on a scale | 19.40 (18.512) | 14.57 (9.049) | 18.43 (15.363) | 20.55 (18.488) | 16.94 (14.256) | 17.96 (15.451)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Treated With Ruxolitinib Cream Who Achieved a ≥ 50% Improvement From Baseline in Facial Assessment of the Vitiligo Area and Severity Index Score (F-VASI50) Compared With Participants Treated With Vehicle at Week 24
Description: An F-VASI50 responder achieved at least 50% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of body surface area [BSA]) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; Week 24
Population: Intent-to-Treat (ITT) Population: all randomized participants. Treatment groups were to be defined according to the treatment assignment at the time of randomization regardless of the actual ruxolitinib cream or vehicle cream participants might have applied during their participation in the study. Missing post-Baseline values were considered as not having achieved responses for visits up to Week 52.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
percentage of participants | 3.1 | 32.3 | 25.8 | 50.0 | 45.5
Statistical Analysis 1: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.15% QD; Test type: Superiority; p = 0.0057, exact logistic regression — The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 13.79, 95% CI 2-sided [1.73 to 640.85]
Statistical Analysis 2: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.5% QD; Test type: Superiority; p = 0.0243, exact logistic regression — The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 10.30, 95% CI 2-sided [1.24 to 487.28]
Statistical Analysis 3: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% QD; Test type: Superiority; p < 0.0001, exact logistic regression — The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 28.48, 95% CI 2-sided [3.74 to 1305.2]
Statistical Analysis 4: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% BID; Test type: Superiority; p = 0.0001, exact logistic regression — The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 24.66, 95% CI 2-sided [3.28 to 1121.4]

2. Secondary Outcome: Percentage of Participants Who Achieved a Facial Assessment of the Physician's Global Vitiligo Assessment (F-PhGVA) of Clear or Almost Clear
Description: The severity of vitiligo was assessed by the physician using the PhGVA, which has a 5-point scale. 0=clear, no signs of vitiligo; 1=almost clear, only specks of depigmentation present; 2=mild disease, pigmented and depigmented areas are equal; 3=moderate disease, more or complete depigmentation (may include < 30% hair whitening); 4=severe disease, complete depigmentation plus > 30% hair whitening.
Time Frame: Week 24
Population: ITT Population. Missing post-Baseline values were considered as not having achieved F-PhGVA response for visits up to Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
percentage of participants | 0 | 3.2 | 9.7 | 13.3 | 9.1
Statistical Analysis 1: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.15% QD; Test type: Superiority; p = 0.4936, exact logistic regression — The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 1.03, 95% CI 2-sided [lower limit 0.05] (The upper limit of the confidence interval was not estimatable because there were too few participants with a response of clear or almost clear.)
Statistical Analysis 2: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.5% QD; Test type: Superiority; p = 0.1140, exact logistic regression — The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 4.16, 95% CI 2-sided [lower limit 0.62] (The upper limit of the confidence interval was not estimatable because there were too few participants with a response of clear or almost clear.)
Statistical Analysis 3: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% QD; Test type: Superiority; p = 0.0501, exact logistic regression — The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 6.10, 95% CI 2-sided [lower limit 1.00] (The upper limit of the confidence interval was not estimatable because there were too few participants with a response of clear or almost clear.)
Statistical Analysis 4: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% BID; Test type: Superiority; p = 0.1257, exact logistic regression — The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 3.89, 95% CI 2-sided [lower limit 0.58] (The upper limit of the confidence interval was not estimatable because there were too few participants with a response of clear or almost clear.)

3. Secondary Outcome: Percentage of Participants Who Achieved a ≥ 50% Improvement From Baseline in Full Body Assessment of Vitiligo Area and Severity Index (T-VASI) at Week 52
Description: T-VASI was measured by the percentage of vitiligo involvement from all body regions (percentage of BSA; assessed by the Investigator) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was derived by multiplying the vitiligo involvement values by the percentage of affected skin for each body site and summing all values (possible range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; Week 52
Population: ITT Population. Missing post-Baseline values were considered as not having achieved responses for visits up to Week 52. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Ruxolitinib Cream 0.15% QD: Ruxolitinib cream 0.15% QD in the morning (vehicle cream in the evening) for 52 weeks (combined vehicle-controlled and continued double-blind periods) in participants who saw greater than or equal to 25% improvement in F-VASI score at Week 24, followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID: Participants who were randomized to the vehicle group and participants who were randomized to ruxolitinib cream 0.15% QD who did not achieve a 25% improvement in F-VASI score at Week 24 who crossed over to ruxolitinib cream 0.5% QD in the morning (vehicle cream in the evening) for 28 weeks (Week 24 to Week 52 [continued double-blind treatment period]), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID: Participants who were randomized to the vehicle group and participants who were randomized to ruxolitinib cream 0.15% QD who did not achieve a 25% improvement in F-VASI score at Week 24 who crossed over to ruxolitinib cream 1.5% QD in the morning (vehicle cream in the evening) for 28 weeks (Week 24 to Week 52 [continued double-blind treatment period]), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID: Participants who were randomized to the vehicle group and participants who were randomized to ruxolitinib cream 0.15% QD who did not achieve a 25% improvement in F-VASI score at Week 24 who crossed over to ruxolitinib cream 1.5% BID for 28 weeks (Week 24 to Week 52 [continued double-blind treatment period]), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Ruxolitinib Cream 0.5% QD: 1.5% BID: Ruxolitinib cream 0.5% QD in the morning (vehicle cream in the evening) for 52 weeks (combined vehicle-controlled and continued double-blind periods), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Ruxolitinib Cream 1.5% QD: 1.5 % BID: Ruxolitinib cream 1.5% QD in the morning (vehicle cream in the evening) for 52 weeks (combined vehicle-controlled and continued double-blind periods), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Ruxolitinib Cream 1.5% BID: 1.5% BID: Ruxolitinib cream 1.5% BID for 52 weeks (combined vehicle-controlled and continued double-blind periods), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 10 | 14 | 12 | 13 | 31 | 30 | 33
percentage of participants | 50 | 21.4 | 16.7 | 15.4 | 25.8 | 30.0 | 36.4
Statistical Analysis 1: Comparison: Ruxolitinib Cream 0.5% QD: 1.5% BID vs Ruxolitinib Cream 1.5% QD: 1.5 % BID; Test type: Superiority; p = 0.9794, exact logistic regression; The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.33 to 4.33]
Statistical Analysis 2: Comparison: Ruxolitinib Cream 0.5% QD: 1.5% BID vs Ruxolitinib Cream 1.5% BID: 1.5% BID; Test type: Superiority; p = 0.4893, exact logistic regression; The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.51 to 5.86]

4. Secondary Outcome: Dose Response on Percentage Change From Baseline in F-VASI
Time Frame: up to 156 weeks
Population: Based on the data for percentage change from Baseline in F-VASI and T-VASI scores during the treatment periods, the Emax model was not appropriate; therefore, the dose responses were not assessed.
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) and Any Grade 3 or Higher TEAE up to Week 24
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. A TEAE was an AE reported for the first time or the worsening of a pre-existing event after first application of study drug. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) v4.03 Grades 1 through 4. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent intervention indicated.
Time Frame: up to 24 weeks
Population: Safety Population: all participants who applied at least 1 dose of study drug. Treatment groups for this population were to be determined according to the actual treatment the participant received on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
Participants
  Any TEAE | 20 | 20 | 22 | 22 | 20
  Any Grade 3 or higher TEAE | 0 | 0 | 0 | 0 | 1

6. Secondary Outcome: Number of Participants With Any TEAE and Any Grade 3 or Higher TEAE up to Week 52
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. A TEAE was an AE reported for the first time or the worsening of a pre-existing event after first application of study drug. The severity of AEs was assessed using CTCAE v4.03 Grades 1 through 4. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent intervention indicated.
Time Frame: up to 52 weeks
Population: Safety Population. Treatment groups for this population were to be determined according to the actual treatment the participant received on Day 1. Analysis from Day 1 to Week 52 was conducted in participants randomized to receive ruxolitinib cream 0.5% QD, ruxolitinib cream 1.5% QD, or ruxolitinib cream 1.5% BID during the vehicle-controlled period (Day 1 to Week 24).
Measure: Count of Participants; unit: Participants
Groups:
- Vehicle/Ruxolitinib Cream 0.15% to 1.5% QD: 1.5% BID: Participants who were randomized to the vehicle group and participants who were randomized to ruxolitinib cream 0.15% QD who did not achieve a 25% improvement in F-VASI score at Week 24 who crossed over to ruxolitinib cream 1.5% QD in the morning (vehicle cream in the evening) for 28 weeks (Week 24 to Week 52 [continued double-blind treatment period]), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
- Vehicle/Ruxolitinib Cream 0.15% to 1.5% BID: 1.5% BID: Participants who were randomized to the vehicle group and participants who were randomized to ruxolitinib cream 0.15% QD who did not achieve a 25% improvement in F-VASI score at Week 24 who crossed over to ruxolitinib cream 1.5% BID for 28 weeks (Week 24 to Week 52 [continued double-blind treatment period]), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 31 | 30 | 33
Participants
  Any TEAE |  |  |  |  | 26 | 23 | 23
  Any Grade 3 or higher TEAE |  |  |  |  | 2 | 1 | 1

7. Secondary Outcome: Number of Participants With Any TEAE and Any Grade 3 or Higher TEAE From Week 24 to Week 52
Description: as for outcome 6
Time Frame: Week 24 to Week 52
Population: Safety Population. Treatment groups for this population were to be determined according to the actual treatment the participant received on Day 1. Analysis was conducted in participants who were randomized to ruxolitinib cream 0.15% QD and vehicle groups in the vehicle-controlled period (Day 1 to Week 24) and then had a dose in the continued double-blind period (Week 24 to Week 52).
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 0 | 0 | 0
Participants
  Any TEAE | 9 | 6 | 5 | 9 |  |  |
  Any Grade 3 or higher TEAE | 0 | 0 | 0 | 0 |  |  |

8. Secondary Outcome: Number of Participants Who Applied Ruxolitinib 1.5% Cream BID Throughout Study Participation With Any TEAE and Any Grade 3 or Higher TEAE
Description: as for outcome 6
Time Frame: up to Week 156
Population: Safety Population. Treatment groups for this population were to be determined according to the actual treatment the participant received on Day 1. Analysis was only conducted in participants who received ruxolitinib cream 1.5% BID on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 33
Participants
  Any TEAE |  |  |  |  |  |  | 26
  Any Grade 3 or higher TEAE |  |  |  |  |  |  | 1

9. Secondary Outcome: Number of Participants With Any TEAE and Any Grade 3 or Higher TEAE From Week 52 to Week 156
Description: as for outcome 6
Time Frame: Week 52 to Week 156
Population: Open-label Evaluable Population: all randomized participants who received at least 1 dose of study drug in the Open-label Period
Measure: Count of Participants; unit: Participants
Groups:
- Ruxolitinib Cream 1.5% QD: 1.5% BID: Ruxolitinib cream 1.5% QD in the morning (vehicle cream in the evening) for 52 weeks (combined vehicle-controlled and continued double-blind periods), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
Arm/Group | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% BID: 1.5% BID | Cross-over
Number analyzed (Participants) | 28 | 21 | 28 | 46
Participants
  Any TEAE | 15 | 16 | 13 | 25
  Any Grade 3 or higher TEAE | 0 | 2 | 0 | 2

10. Secondary Outcome: Mean Change From Baseline in F-VASI Score at Week 24
Description: F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed. Mixed-model for Repeated Measures (MMRM) model for post-Baseline measures: (response variable = treatment + stratification factor [age ≤30 versus >30] + visit + treatment*visit). All post-Baseline visits up to Week 24 were included in the model.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
scores on a scale | 0.05 (0.11) | -0.39 (0.11) | -0.35 (0.11) | -0.63 (0.11) | -0.46 (0.10)
Statistical Analysis 1: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.15% QD; Test type: Superiority; p = 0.0056, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; Least squares mean (LSM) difference = -0.44, 95% CI 2-sided [-0.75 to -0.13], Standard Error of Mean 0.16 — LSM difference = treatment minus vehicle
Statistical Analysis 2: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.5% QD; Test type: Superiority; p = 0.0095, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -0.40, 95% CI 2-sided [-0.70 to -0.10], Standard Error of Mean 0.15 — LSM difference = treatment minus vehicle
Statistical Analysis 3: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% QD; Test type: Superiority; p < 0.0001, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -0.68, 95% CI 2-sided [-0.99 to -0.37], Standard Error of Mean 0.16 — LSM difference = treatment minus vehicle
Statistical Analysis 4: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% BID; Test type: Superiority; p = 0.0011, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -0.51, 95% CI 2-sided [-0.80 to -0.21], Standard Error of Mean 0.15 — LSM difference = treatment minus vehicle

11. Secondary Outcome: Mean Change From Baseline in F-VASI Score at Weeks 52, 104, and 156
Description: as for outcome 10
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
scores on a scale
  Baseline | 0.77 (0.387) | 1.21 (0.891) | 1.66 (0.993) | 1.14 (0.714) | 1.22 (0.705) | 1.45 (0.980) | 1.26 (0.808)
  Change from Baseline at Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Change from Baseline at Week 52 | -0.59 (0.459) | -0.67 (0.811) | -1.02 (1.058) | -0.58 (0.783) | -0.58 (0.578) | -0.74 (0.797) | -0.76 (0.610)
  Change from Baseline at Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Change from Baseline at Week 104 | -0.66 (0.444) | -0.97 (1.061) | -1.79 (1.077) | -0.87 (0.903) | -1.00 (0.697) | -1.17 (0.961) | -0.99 (0.817)
  Change from Baseline at Week 156: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Change from Baseline at Week 156 | -0.66 (0.124) | -0.98 (1.092) | -1.40 (1.018) | -0.65 (0.557) | -0.71 (0.490) | -0.95 (0.949) | -1.23 (0.887)

12. Secondary Outcome: Percentage Change From Baseline in F-VASI Score at Week 24
Description: F-VASI was measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement). Percentage change = ([post-Baseline value minus Baseline value]/Baseline value) X 100.
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed. MMRM model for post-Baseline measures: (response variable = treatment + stratification factor [age ≤30 versus >30] + visit + treatment*visit). All post-Baseline visits up to Week 24 were included in the model.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
percent change | 6.02 (7.23) | -30.69 (7.39) | -29.10 (6.93) | -40.00 (7.39) | -37.78 (6.89)
Statistical Analysis 1: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.15% QD; Test type: Superiority; p = 0.0005, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -36.71, 95% CI 2-sided [-57.15 to -16.27], Standard Error of Mean 10.34 — LSM difference = treatment minus vehicle
Statistical Analysis 2: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.5% QD; Test type: Superiority; p = 0.0006, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LM difference = -35.12, 95% CI 2-sided [-54.91 to -15.33], Standard Error of Mean 10.01 — LSM difference = treatment minus vehicle
Statistical Analysis 3: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% QD; Test type: Superiority; p < 0.0001, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -46.02, 95% CI 2-sided [-66.47 to -25.57], Standard Error of Mean 10.35 — LSM difference = treatment minus vehicle
Statistical Analysis 4: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% BID; Test type: Superiority; p < 0.0001, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -43.80, 95% CI 2-sided [-63.52 to -24.07], Standard Error of Mean 9.98 — LSM difference = treatment minus vehicle

13. Secondary Outcome: Percentage Change From Baseline in F-VASI Score at Weeks 52, 104, and 156
Description: as for outcome 12
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percent change
  Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52 | -72.21 (26.837) | -50.60 (34.954) | -52.43 (36.412) | -40.79 (37.082) | -45.54 (35.148) | -55.63 (42.823) | -57.34 (50.115)
  Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104 | -77.67 (22.974) | -71.12 (31.087) | -82.87 (32.756) | -60.28 (64.708) | -74.89 (25.524) | -77.76 (24.086) | -78.78 (28.400)
  Week 156: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156 | -87.95 (8.207) | -66.83 (45.106) | -91.25 (14.631) | -59.16 (42.627) | -76.25 (20.126) | -76.76 (23.924) | -89.52 (14.899)

14. Secondary Outcome: Percentage of Participants Who Achieved an F-VASI50 at Weeks 52, 104, and 156
Description: An F-VASI50 responder achieved at least 50% improvement from Baseline in F-VASI, measured by the percentage of vitiligo involvement (percentage of BSA) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment), or 100% (no pigment). The percentage of BSA (hand unit) vitiligo involvement was estimated to the nearest 0.1% by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate the percentage of BSA vitiligo involvement. F-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site on the face and summing the values of all sites (possible range: 0-3; lower scores indicate increased improvement).
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percentage of participants
  Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 31 | 30 | 33
  Week 52 | 90.0 | 64.3 | 50.0 | 38.5 | 45.2 | 43.3 | 57.6
  Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104 | 88.9 | 87.5 | 88.9 | 77.8 | 78.9 | 83.3 | 89.5
  Week 156: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156 | 100.0 | 75.0 | 100.0 | 60.0 | 87.5 | 87.5 | 100.0

15. Secondary Outcome: Percentage Change From Baseline in F-BSA Repigmentation at Week 24
Description: F-BSA involvement was the proportion of the facial body surface area with vitiligo. The area "Face" was defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically and laterally from the corner of the mouth to the tragus. The area "Face" did not include the surface area of the lips, scalp, ears, or neck, but included the nose and eyelids. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-Baseline value minus Baseline value]/Baseline value) X 100.
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
percent change | 6.49 (32.028) | -19.82 (24.928) | -17.55 (25.453) | -19.53 (38.612) | -27.76 (30.996)

16. Secondary Outcome: Percentage Change From Baseline in F-BSA Repigmentation at Weeks 52, 104, and 156
Description: as for outcome 15
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percent change
  Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52 | -55.18 (36.091) | -37.94 (32.569) | -33.39 (40.095) | -15.64 (29.733) | -34.67 (37.769) | -38.37 (38.660) | -44.29 (35.253)
  Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104 | -42.86 (31.282) | -67.61 (29.683) | -76.57 (31.260) | -45.65 (59.599) | -54.49 (34.411) | -63.56 (28.543) | -59.49 (38.186)
  Week 156: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156 | -33.04 (6.313) | -59.17 (40.586) | -90.50 (16.240) | -16.89 (56.706) | -55.80 (33.310) | -59.58 (27.106) | -72.58 (31.024)

17. Secondary Outcome: Percentage Change From Baseline in T-BSA Repigmentation at Week 24
Description: T-BSA involvement was the proportion of the body surface area with vitiligo. Body surface area assessment was performed by the Palmar Method. Body surface area was estimated to the nearest 0.1%. The approximate size of the participant's entire palmar surface (i.e., the palm plus 5 digits) was considered as 1% BSA, and the approximate size of the participant's thumb was considered as 0.1% BSA. Percentage change = ([post-Baseline value minus Baseline value]/Baseline value) X 100.
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
percent change | 3.35 (8.314) | -13.97 (25.396) | -10.83 (15.646) | -17.19 (22.490) | -13.60 (20.443)

18. Secondary Outcome: Percentage Change From Baseline in T-BSA Repigmentation at Weeks 52, 104, and 156
Description: as for outcome 17
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percent change
  Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52 | -39.53 (32.599) | -8.72 (26.010) | -2.72 (23.014) | -8.73 (21.630) | -15.13 (21.296) | -27.33 (27.568) | -27.59 (26.770)
  Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104 | -42.42 (32.208) | -30.49 (36.289) | -30.08 (30.717) | -21.08 (30.323) | -33.19 (30.127) | -33.94 (26.573) | -32.46 (33.190)
  Week 156: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156 | -59.44 (51.920) | -46.58 (30.723) | -34.93 (35.391) | -37.95 (23.651) | -29.59 (32.261) | -10.55 (53.863) | -46.88 (19.304)

19. Secondary Outcome: Mean Change From Baseline in T-VASI Score at Week 24
Description: T-VASI was calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement). Change from Baseline (BL) was calculated as the post-BL value minus the BL value.
Time Frame: Baseline; Week 24
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
scores on a scale | 0.57 (0.92) | -2.27 (0.94) | -2.18 (0.88) | -4.51 (0.94) | -3.52 (0.87)
Statistical Analysis 1: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.15% QD; Test type: Superiority; p = 0.0326, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -2.84, 95% CI 2-sided [-5.44 to -0.24], Standard Error of Mean 1.32 — LSM difference = treatment minus vehicle
Statistical Analysis 2: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.5% QD; Test type: Superiority; p = 0.0333, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -2.74, 95% CI 2-sided [-5.26 to -0.22], Standard Error of Mean 1.28 — LSM difference = treatment minus vehicle
Statistical Analysis 3: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% QD; Test type: Superiority; p = 0.0002, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -5.08, 95% CI 2-sided [-7.68 to -2.48], Standard Error of Mean 1.31 — LSM difference = treatment minus vehicle
Statistical Analysis 4: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% BID; Test type: Superiority; p = 0.0016, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -4.08, 95% CI 2-sided [-6.59 to -1.57], Standard Error of Mean 1.27 — LSM difference = treatment minus vehicle

20. Secondary Outcome: Mean Change From Baseline in T-VASI Score at Weeks 52, 104, and 156
Description: T-VASI was calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement). Change from BL was calculated as the post-BL value minus the BL value.
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
scores on a scale
  Baseline | 9.56 (7.090) | 13.47 (11.655) | 22.82 (19.187) | 20.75 (15.973) | 18.43 (15.363) | 20.55 (18.488) | 16.94 (14.256)
  Change from Baseline at Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Change from Baseline at Week 52 | -4.59 (4.979) | -2.88 (2.934) | -3.21 (4.536) | -3.88 (5.642) | -3.97 (6.284) | -7.37 (7.403) | -6.14 (7.442)
  Change from Baseline at Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Change from Baseline at Week 104 | -6.02 (5.476) | -5.32 (5.615) | -9.71 (9.398) | -6.62 (7.054) | -7.19 (9.079) | -10.77 (9.658) | -7.74 (5.927)
  Change from Baseline at Week 156: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Change from Baseline at Week 156 | -2.33 (0.269) | -10.23 (13.533) | -11.31 (12.185) | -7.82 (4.209) | -4.72 (3.622) | -7.02 (9.577) | -8.77 (4.996)

21. Secondary Outcome: Percentage Change From Baseline in T-VASI Score at Week 24
Description: T-VASI was calculated with contributions from 6 sites. The percentage of vitiligo involvement was estimated in hand units (percentage of BSA estimated to nearest 0.1%) by the Investigator using the Palmar Method. The Investigator used his/her hand to mimic the participant's hand size to evaluate percent BSA vitiligo involvement. The degree of depigmentation for each site was estimated to the nearest percentage: 0% (no depigmentation present), 10% (only specks of depigmentation present), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each site and summing the values (range: 0-100; lower scores indicate increased improvement).
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed. Percentage change = ([post-Baseline value minus Baseline value]/Baseline value) X 100. MMRM model for post-Baseline measures: (response variable = treatment + stratification factor [age ≤30 versus >30] + visit + treatment*visit). All post-Baseline visits up to Week 24 were included in the model.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
percent change | 2.65 (4.89) | -20.88 (5.00) | -15.82 (4.69) | -27.16 (4.99) | -22.91 (4.65)
Statistical Analysis 1: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.15% QD; Test type: Superiority; p = 0.0010, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -23.53, 95% CI 2-sided [-37.35 to -9.71], Standard Error of Mean 6.99 — LSM difference = treatment minus vehicle
Statistical Analysis 2: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.5% QD; Test type: Superiority; p = 0.0072, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -18.47, 95% CI 2-sided [-31.86 to -5.08], Standard Error of Mean 6.77 — LSM difference = treatment minus vehicle
Statistical Analysis 3: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% QD; Test type: Superiority; p < 0.0001, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -29.81, 95% CI 2-sided [-43.61 to -16.00], Standard Error of Mean 6.98 — LSM difference = treatment minus vehicle
Statistical Analysis 4: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% BID; Test type: Superiority; p = 0.0002, Log Rank; Treatment comparisons were performed using the log-rank test stratified by randomization stratification factor; LSM difference = -25.56, 95% CI 2-sided [-38.89 to -12.22], Standard Error of Mean 6.75 — LSM difference = treatment minus vehicle

22. Secondary Outcome: Percentage Change From Baseline in T-VASI Score at Weeks 52, 104, and 156
Description: as for outcome 21
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed. Percentage change = ([post-Baseline value minus Baseline value]/Baseline value) X 100.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percent change
  Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52 | -50.71 (33.310) | -25.12 (31.556) | -19.75 (26.484) | -20.00 (29.264) | -24.67 (29.649) | -41.90 (35.865) | -41.67 (26.451)
  Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104 | -60.96 (32.259) | -49.35 (39.319) | -49.07 (29.091) | -38.70 (38.663) | -46.44 (31.668) | -52.14 (33.559) | -50.03 (26.905)
  Week 156: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156 | -71.10 (31.448) | -59.33 (40.055) | -47.31 (34.610) | -49.96 (27.555) | -44.69 (30.718) | -14.97 (58.982) | -62.80 (20.904)

23. Secondary Outcome: Mean Change From Baseline in Vitiligo European Task Force (VETF) Scale Scores at Week 24: Total Spreading
Description: The VETF-proposed system combines analysis of extent (0%-100% BSA), stage of disease (staging), and disease progression (spreading); each component is evaluated and reported independently. Staging is based on cutaneous and hair pigmentation in vitiligo patches. Disease is staged 0 to 4 on the largest macule in each of 5 body regions, except hands and feet, which are assessed separately and globally as 1 unique area. Stage 0=normal pigmentation, Stage 1=incomplete pigmentation, Stage 2=complete depigmentation (a few white hairs do not change stage), Stage 3=partial hair whitening (<30%), Stage 4=complete hair whitening; total score of 0 (less severe disease) to 20 (more severe disease). Disease progression is based on assessing the largest patch in each of 5 body areas: -1=regressive vitiligo (ongoing subclinical repigmentation), 0=similar limits, 1=progressive vitiligo (ongoing subclinical depigmentation); total score of -5 (improving disease) to +5 (more severe disease spread).
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
scores on a scale
  Baseline | 1.78 (2.166) | 2.74 (2.422) | 1.84 (2.238) | 1.83 (2.102) | 1.21 (2.233)
  Change from Baseline at Week 24: number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
  Change from Baseline at Week 24 | -1.12 (2.566) | -3.15 (3.246) | -3.27 (3.532) | -3.12 (2.971) | -3.58 (3.042)

24. Secondary Outcome: Mean Change From Baseline in VETF Scale Scores at Weeks 52 and 104: Total Spreading
Description: as for outcome 23
Time Frame: Baseline; Weeks 52 and 104
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
scores on a scale
  Baseline | 2.73 (2.328) | 2.43 (2.277) | 1.21 (2.607) | 2.21 (1.968) | 1.84 (2.238) | 1.83 (2.102) | 1.21 (2.233)
  Change from Baseline at Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Change from Baseline at Week 52 | -4.70 (3.683) | -4.14 (3.592) | -3.83 (3.538) | -3.85 (3.211) | -3.48 (3.622) | -3.86 (3.395) | -3.66 (2.742)
  Change from Baseline at Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Change from Baseline at Week 104 | -5.00 (4.153) | -4.25 (3.196) | -4.22 (3.667) | -5.11 (3.371) | -3.16 (3.516) | -3.56 (3.034) | -3.26 (3.034)

25. Secondary Outcome: Mean Change From Baseline in VETF Scale Scores at Week 24: Total Percentage Area
Description: as for outcome 23
Time Frame: Baseline; Week 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
scores on a scale
  Baseline | 22.81 (20.843) | 16.26 (11.006) | 22.35 (20.878) | 24.63 (22.236) | 20.79 (16.192)
  Change from Baseline at Week 24: number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
  Change from Baseline at Week 24 | 0.38 (1.329) | -1.08 (3.867) | -2.43 (4.797) | -3.27 (6.744) | -2.71 (4.591)

26. Secondary Outcome: Mean Change From Baseline in VETF Scale Scores at Weeks 52 and 104: Total Percentage Area
Description: as for outcome 23
Time Frame: Baseline; Weeks 52 and 104
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
scores on a scale
  Baseline | 9.18 (6.509) | 16.43 (11.979) | 24.50 (21.841) | 24.50 (18.798) | 22.35 (20.878) | 24.63 (22.236) | 20.79 (16.192)
  Change from Baseline at Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Change from Baseline at Week 52 | -3.10 (3.814) | -1.86 (2.905) | -1.17 (3.486) | -1.92 (6.211) | -3.93 (7.191) | -5.71 (8.463) | -4.48 (6.127)
  Change from Baseline at Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Change from Baseline at Week 104 | -3.89 (4.226) | -4.75 (5.994) | -5.11 (4.226) | -4.44 (7.367) | -8.00 (10.392) | -7.78 (8.695) | -6.26 (6.682)

27. Secondary Outcome: Percentage Change From Baseline in VETF Scale Scores at Week 24: Total Percentage Area
Description: as for outcome 23
Time Frame: Baseline; Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
percent change | 2.61 (9.497) | -10.61 (29.408) | -13.87 (25.296) | -14.09 (20.321) | -13.10 (17.605)

28. Secondary Outcome: Percentage Change From Baseline in VETF Scale Scores at Weeks 52 and 104: Total Percentage Area
Description: as for outcome 23
Time Frame: Baseline; Weeks 52 and 104
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percent change
  Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52 | -32.01 (35.629) | -7.39 (21.571) | -10.57 (22.300) | -7.13 (25.967) | -19.73 (30.730) | -22.36 (23.593) | -25.41 (24.049)
  Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104 | -39.30 (37.071) | -23.05 (29.233) | -34.03 (27.992) | -18.49 (36.527) | -35.55 (34.039) | -30.40 (22.940) | -29.19 (39.767)

29. Secondary Outcome: Mean Change From Baseline in VETF Scale Scores at Week 24: Total Staging
Description: as for outcome 23
Time Frame: Baseline; Week 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Ruxolitinib Cream 1.5% QD: Ruxolitinib cream 1.5% QD Ruxolitinib cream 1.5% QD in the morning (vehicle cream in the evening) for 52 weeks (combined vehicle-controlled and continued double-blind periods), followed by ruxolitinib cream 1.5% BID in a 104-week open-label extension period.
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
scores on a scale
  Baseline | 10.03 (3.515) | 9.29 (3.013) | 10.03 (3.945) | 9.97 (3.000) | 8.42 (3.464)
  Change from Baseline at Week 24: number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
  Change from Baseline at Week 24 | -1.15 (3.184) | -1.62 (2.282) | -1.57 (2.687) | -1.96 (3.561) | -0.74 (2.633)

30. Secondary Outcome: Mean Change From Baseline in VETF Scale Scores at Weeks 52 and 104: Total Staging
Description: as for outcome 23
Time Frame: Baseline; Weeks 52 and 104
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
scores on a scale
  Baseline | 8.64 (2.908) | 8.43 (2.901) | 11.29 (2.128) | 10.07 (3.668) | 10.03 (3.945) | 9.97 (3.000) | 8.42 (3.464)
  Change from Baseline at Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Change from Baseline at Week 52 | -3.10 (3.247) | -1.29 (2.301) | -2.17 (3.157) | -2.62 (2.844) | -2.41 (3.030) | -3.48 (2.960) | -1.38 (2.555)
  Change from Baseline at Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Change from Baseline at Week 104 | -3.44 (3.358) | -2.75 (3.694) | -2.22 (3.866) | -2.89 (1.537) | -2.84 (2.754) | -4.00 (3.049) | -1.68 (2.730)

31. Secondary Outcome: Percentage Change From Baseline in VETF Scale Scores at Week 24: Total Staging
Description: as for outcome 23
Time Frame: Baseline; Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
percent change | -7.58 (18.740) | -17.52 (22.267) | -13.55 (21.200) | -17.00 (31.798) | -4.46 (38.916)

32. Secondary Outcome: Percentage Change From Baseline in VETF Scale Scores at Weeks 52 and 104: Total Staging
Description: as for outcome 23
Time Frame: Baseline; Weeks 52 and 104
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percent change
  Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52 | -33.48 (25.022) | -12.70 (24.012) | -17.31 (22.623) | -23.88 (19.262) | -21.45 (24.571) | -30.00 (22.563) | -12.99 (29.585)
  Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104 | -37.20 (29.132) | -24.29 (30.439) | -16.55 (27.268) | -32.06 (12.311) | -27.76 (23.202) | -35.20 (23.904) | -14.09 (26.969)

33. Secondary Outcome: Percentage of Participants in Each Facial Assessment of the Physician's Global Vitiligo Assessment (F-PhGVA) Category at Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
percentage of participants
  0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  1 | 0.0 | 3.2 | 9.7 | 13.3 | 9.1
  2 | 6.3 | 16.1 | 16.1 | 20.0 | 27.3
  3 | 40.6 | 64.5 | 61.3 | 36.7 | 54.5
  4 | 34.4 | 0.0 | 9.7 | 16.7 | 3.0
  Missing at the visit | 18.8 | 16.1 | 3.2 | 13.3 | 6.1
Statistical Analysis 1: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.15% QD; Test type: Superiority; p = 0.4936, exact logistic regression; The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 1.03, 95% CI 2-sided [lower limit 0.05] (The upper limit of the confidence interval was not estimatable because there were too few participants with a response of clear or almost clear.)
Statistical Analysis 2: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 0.5% QD; Test type: Superiority; p = 0.1140, exact logistic regression; The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 4.16, 95% CI 2-sided [lower limit 0.62] (The upper limit of the confidence interval was not estimatable because there were too few participants with a response of clear or almost clear.)
Statistical Analysis 3: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% QD; Test type: Superiority; p = 0.0501, exact logistic regression; The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 6.10, 95% CI 2-sided [lower limit 1.00] (The upper limit of the confidence interval was not estimatable because there were too few participants with a response of clear or almost clear.)
Statistical Analysis 4: Comparison: Vehicle Twice Daily (BID) vs Ruxolitinib Cream 1.5% BID; Test type: Superiority; p = 0.1257, exact logistic regression; The exact logistic regression model includes treatment and stratification factor (age ≤30 versus >30); Odds Ratio (OR) = 3.89, 95% CI 2-sided [lower limit 0.58] (The upper limit of the confidence interval was not estimatable because there were too few participants with a response of clear or almost clear.)

34. Secondary Outcome: Percentage of Participants in Each Facial Assessment of the PhGVA (F-PhGVA) Category at Weeks 52, 104 and 156
Description: as for outcome 2
Time Frame: Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percentage of participants
  Week 52, 0: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.9 | 4.8 | 0.0
  Week 52, 1: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 1 | 20.0 | 14.3 | 8.3 | 7.7 | 10.3 | 14.3 | 24.1
  Week 52, 2: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 2 | 60.0 | 7.1 | 33.3 | 46.2 | 17.2 | 28.6 | 37.9
  Week 52, 3: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 3 | 20.0 | 71.4 | 50.0 | 46.2 | 55.2 | 42.9 | 31.0
  Week 52, 4: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 4 | 0.0 | 7.1 | 8.3 | 0.0 | 10.3 | 9.5 | 6.9
  Week 104, 0: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 0 | 0.0 | 0.0 | 11.1 | 11.1 | 5.3 | 11.1 | 15.8
  Week 104, 1: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 1 | 55.6 | 50.0 | 33.3 | 22.2 | 31.6 | 33.3 | 31.6
  Week 104, 2: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 2 | 33.3 | 25.0 | 33.3 | 22.2 | 36.8 | 27.8 | 26.3
  Week 104, 3: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 3 | 11.1 | 25.0 | 11.1 | 44.4 | 26.3 | 27.8 | 21.1
  Week 104, 4: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 4 | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 0.0 | 5.3
  Week 156, 0: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 0 | 0.0 | 0.0 | 60.0 | 0.0 | 25.0 | 0.0 | 33.3
  Week 156, 1: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 1 | 0.0 | 50.0 | 0.0 | 60.0 | 12.5 | 37.5 | 55.6
  Week 156, 2: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 2 | 100.0 | 0.0 | 20.0 | 20.0 | 50.0 | 25.0 | 0.0
  Week 156, 3: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 3 | 0.0 | 50.0 | 20.0 | 20.0 | 12.5 | 37.5 | 11.1
  Week 156, 4: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

35. Secondary Outcome: Percentage of Participants in Each Total Body Assessment of the PhGVA (T-PhGVA) Category at Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 26 | 26 | 30 | 26 | 31
percentage of participants
  0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  1 | 0.0 | 0.0 | 3.3 | 0.0 | 3.2
  2 | 11.5 | 23.1 | 20.0 | 23.1 | 35.5
  3 | 57.7 | 76.9 | 70.0 | 61.5 | 58.1
  4 | 30.8 | 0.0 | 6.7 | 15.4 | 3.2

36. Secondary Outcome: Percentage of Participants in Each Total Body Assessment of the PhGVA (T-PhGVA) Category at Weeks 52, 104 and 156
Description: as for outcome 2
Time Frame: Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percentage of participants
  Week 52, 0: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 52, 1: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 1 | 10.0 | 0.0 | 0.0 | 0.0 | 10.3 | 0.0 | 6.9
  Week 52, 2: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 2 | 50.0 | 35.7 | 8.3 | 7.7 | 13.8 | 28.6 | 55.2
  Week 52, 3: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 3 | 40.0 | 57.1 | 83.3 | 84.6 | 69.0 | 61.9 | 31.0
  Week 52, 4: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 4 | 0.0 | 7.1 | 8.3 | 7.7 | 6.9 | 9.5 | 6.9
  Week 104, 0: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 104, 1: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 1 | 0.0 | 25.0 | 11.1 | 11.1 | 5.3 | 0.0 | 0.0
  Week 104, 2: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 2 | 77.8 | 37.5 | 33.3 | 33.3 | 68.4 | 55.6 | 63.2
  Week 104, 3: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 3 | 22.2 | 37.5 | 44.4 | 55.6 | 26.3 | 27.8 | 36.8
  Week 104, 4: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 4 | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 16.7 | 0.0
  Week 156, 0: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 156, 1: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 1 | 50.0 | 50.0 | 20.0 | 0.0 | 25.0 | 0.0 | 11.1
  Week 156, 2: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 2 | 50.0 | 0.0 | 0.0 | 60.0 | 50.0 | 62.5 | 66.7
  Week 156, 3: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 3 | 0.0 | 50.0 | 60.0 | 40.0 | 25.0 | 25.0 | 22.2
  Week 156, 4: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 4 | 0.0 | 0.0 | 20.0 | 0.0 | 0.0 | 12.5 | 0.0

37. Secondary Outcome: Percentage of Participants in Each Facial Assessment of the Patient's Global Vitiligo Assessment (F-PaGVA) Category at Week 24
Description: The severity of vitiligo was assessed by the participant using the PaGVA, which has a 5-point scale. The participant was asked the following: How severe is your vitiligo on your face (or total body) with respect to the area covered by white skin? Responses: 0=no white patches (no vitiligo); 1=mild; 2=moderate; 3=severe; 4=very severe.
Time Frame: Week 24
Population: ITT Population. Missing post-Baseline values were considered as not having achieved F-PaGVA response for visits up to Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
percentage of participants
  0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  1 | 9.4 | 16.1 | 12.9 | 16.7 | 33.3
  2 | 31.3 | 38.7 | 41.9 | 40.0 | 27.3
  3 | 28.1 | 25.8 | 35.5 | 20.0 | 24.2
  4 | 15.6 | 3.2 | 6.5 | 10.0 | 9.1
  Missing at the visit | 15.6 | 16.1 | 3.2 | 13.3 | 6.1

38. Secondary Outcome: Percentage of Participants in Each Facial Assessment of the PaGVA (F-PaGVA) Category at Weeks 52, 104, and 156
Description: as for outcome 37
Time Frame: Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percentage of participants
  Week 52, 0: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.4
  Week 52, 1: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 1 | 50.0 | 21.4 | 16.7 | 30.8 | 24.1 | 30.0 | 44.8
  Week 52, 2: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 2 | 40.0 | 28.6 | 83.3 | 46.2 | 37.9 | 30.0 | 24.1
  Week 52, 3: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 3 | 10.0 | 50.0 | 0.0 | 23.1 | 34.5 | 30.0 | 20.7
  Week 52, 4: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 4 | 0.0 | 0.0 | 0.0 | 0.0 | 3.4 | 10.0 | 6.9
  Week 104, 0: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 5.3 | 5.6 | 5.3
  Week 104, 1: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 1 | 66.7 | 50.0 | 22.2 | 55.6 | 42.1 | 44.4 | 36.8
  Week 104, 2: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 2 | 22.2 | 37.5 | 55.6 | 33.3 | 36.8 | 16.7 | 47.4
  Week 104, 3: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 3 | 11.1 | 12.5 | 22.0 | 11.1 | 15.8 | 22.2 | 5.3
  Week 104, 4: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 11.1 | 5.3
  Week 156, 0: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 0 | 0.0 | 0.0 | 20.0 | 0.0 | 12.5 | 0.0 | 11.1
  Week 156, 1: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 1 | 50.0 | 50.0 | 0.0 | 80.0 | 37.5 | 37.5 | 44.4
  Week 156, 2: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 2 | 50.0 | 50.0 | 80.0 | 20.0 | 50.0 | 50.0 | 22.2
  Week 156, 3: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 11.1
  Week 156, 4: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 11.1

39. Secondary Outcome: Percentage of Participants in Each Total Body Assessment of the PaGVA (T-PaGVA) Category at Week 24
Description: as for outcome 37
Time Frame: Week 24
Population: ITT Population. Missing post-Baseline values were considered as not having achieved T-PaGVA response for visits up to Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
percentage of participants
  0 | 0.0 | 0.0 | 3.2 | 0.0 | 0.0
  1 | 6.3 | 12.9 | 9.7 | 16.7 | 15.2
  2 | 37.5 | 35.5 | 38.7 | 33.3 | 45.5
  3 | 31.3 | 29.0 | 35.5 | 30.0 | 21.2
  4 | 9.4 | 6.5 | 9.7 | 6.7 | 12.1
  Missing at the visit | 15.6 | 16.1 | 3.2 | 13.3 | 6.1

40. Secondary Outcome: Percentage of Participants in Each Total Body Assessment of the PaGVA (T-PaGVA) Category at Weeks 52, 104, and 156
Description: as for outcome 37
Time Frame: Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percentage of participants
  Week 52, 0: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 52, 1: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 1 | 20.0 | 7.1 | 8.3 | 0.0 | 13.8 | 25.0 | 13.8
  Week 52, 2: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 2 | 60.0 | 50.0 | 41.7 | 69.2 | 48.3 | 40.0 | 62.1
  Week 52, 3: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 20 | 29
  Week 52, 3 | 20.0 | 42.9 | 50.0 | 23.1 | 27.6 | 25.0 | 10.3
  Week 52, 4: number analyzed (Participants) | 10 | 14 | 12 | 13 | 20 | 29 | 20
  Week 52, 4 | 0.0 | 0.0 | 0.0 | 7.7 | 10.3 | 10.0 | 13.8
  Week 104, 0: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 104, 1: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 1 | 33.3 | 25.0 | 0.0 | 0.0 | 36.8 | 22.2 | 15.8
  Week 104, 2: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 2 | 55.6 | 50.0 | 44.4 | 77.8 | 42.1 | 44.4 | 57.9
  Week 104, 3: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 3 | 11.1 | 25.0 | 55.6 | 22.2 | 15.8 | 16.7 | 21.1
  Week 104, 4: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 4 | 0.0 | 0.0 | 0.0 | 0.0 | 5.3 | 16.7 | 5.3
  Week 156, 0: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 156, 1: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 1 | 50.0 | 25.0 | 20.0 | 20.0 | 37.5 | 12.5 | 33.3
  Week 156, 2: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 2 | 50.0 | 75.0 | 40.0 | 40.0 | 50.0 | 37.5 | 55.6
  Week 156, 3: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 3 | 0.0 | 0.0 | 40.0 | 40.0 | 12.5 | 25.0 | 0.0
  Week 156, 4: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 25.0 | 11.1

41. Secondary Outcome: Percentage of Participants in Each Patient Global Impression of Change for Vitiligo (PaGIC-V) Category at Week 24
Description: The PaGIC-V is an assessment of improvement by the participant. It is a 7-point scale comparing the vitiligo areas at Baseline with the participant's treated areas of vitiligo at the study visit. The participant answered the following: "Since the start of the treatment you've received in this study, your vitiligo in areas treated with the study drug is: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; and 7, very much worse.
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 27 | 26 | 30 | 26 | 31
percentage of participants
  1 | 7.4 | 3.8 | 6.7 | 11.5 | 6.5
  2 | 0.0 | 19.2 | 13.3 | 19.2 | 22.6
  3 | 22.2 | 34.6 | 50.0 | 53.8 | 35.5
  4 | 37.0 | 26.9 | 23.3 | 11.5 | 25.8
  5 | 22.2 | 11.5 | 6.7 | 0.0 | 9.7
  6 | 11.1 | 3.8 | 0.0 | 3.8 | 0.0
  7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

42. Secondary Outcome: Percentage of Participants in Each PaGIC-V Category at Weeks 52, 104, and 156
Description: as for outcome 41
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percentage of participants
  Week 52, 1: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 1 | 0.0 | 7.1 | 8.3 | 7.7 | 10.3 | 4.8 | 13.8
  Week 52, 2: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 2 | 30.0 | 14.3 | 25.0 | 23.1 | 20.7 | 47.6 | 31.0
  Week 52, 3: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 3 | 30.0 | 42.9 | 58.3 | 46.2 | 55.2 | 38.1 | 27.6
  Week 52, 4: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 4 | 20.0 | 7.1 | 8.3 | 15.4 | 6.9 | 9.5 | 20.7
  Week 52, 5: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 5 | 20.0 | 28.6 | 0.0 | 7.7 | 3.4 | 0.0 | 6.9
  Week 52, 6: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 6 | 0.0 | 0.0 | 0.0 | 0.0 | 3.4 | 0.0 | 0.0
  Week 52, 7: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52, 7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 104, 1: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 1 | 11.1 | 25.0 | 11.1 | 22.2 | 10.5 | 22.2 | 21.1
  Week 104, 2: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 2 | 33.3 | 12.5 | 44.4 | 33.3 | 36.8 | 38.9 | 36.8
  Week 104, 3: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 3 | 22.2 | 62.5 | 33.3 | 22.2 | 47.4 | 22.2 | 36.8
  Week 104, 4: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 4 | 22.2 | 0.0 | 11.1 | 22.2 | 5.3 | 11.1 | 0.0
  Week 104, 5: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 5 | 11.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 5.3
  Week 104, 6: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 6 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 5.6 | 0.0
  Week 104, 7: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104, 7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Week 156, 1: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 1 | 50.0 | 25.0 | 20.0 | 20.0 | 12.5 | 12.5 | 11.1
  Week 156, 2: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 2 | 50.0 | 25.0 | 20.0 | 60.0 | 25.0 | 50.0 | 77.8
  Week 156, 3: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 3 | 0.0 | 50.0 | 40.0 | 0.0 | 62.5 | 12.5 | 11.1
  Week 156, 4: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 4 | 0.0 | 0.0 | 20.0 | 20.0 | 0.0 | 0.0 | 0.0
  Week 156, 5: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0
  Week 156, 6: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 6 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0
  Week 156, 7: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156, 7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

43. Secondary Outcome: Percentage of Participants Who Report a PaGIC-V Score of Very Much Improved or Much Improved at Week 24
Description: as for outcome 41
Time Frame: Baseline; Week 24
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 27 | 26 | 30 | 26 | 31
percentage of participants | 7.4 | 23.1 | 20.0 | 30.8 | 29.0

44. Secondary Outcome: Percentage of Participants Who Report a PaGIC-V Score of Very Much Improved or Much Improved at Weeks 52, 104, and 156
Description: as for outcome 41
Time Frame: Baseline; Weeks 52, 104, and 156
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Cream 0.15% QD | Vehicle/Ruxolitinib Cream 0.15% QD to 0.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% QD: 1.5% BID | Vehicle/Ruxolitinib Cream 0.15% QD to 1.5% BID: 1.5% BID | Ruxolitinib Cream 0.5% QD: 1.5% BID | Ruxolitinib Cream 1.5% QD: 1.5 % BID | Ruxolitinib Cream 1.5% BID: 1.5% BID
Number analyzed (Participants) | 11 | 14 | 14 | 14 | 31 | 30 | 33
percentage of participants
  Week 52: number analyzed (Participants) | 10 | 14 | 12 | 13 | 29 | 21 | 29
  Week 52 | 30.0 | 21.4 | 33.3 | 30.8 | 31.0 | 52.4 | 44.8
  Week 104: number analyzed (Participants) | 9 | 8 | 9 | 9 | 19 | 18 | 19
  Week 104 | 44.4 | 37.5 | 55.6 | 55.6 | 47.4 | 61.1 | 57.9
  Week 156: number analyzed (Participants) | 2 | 4 | 5 | 5 | 8 | 8 | 9
  Week 156 | 100.0 | 50.0 | 40.0 | 80.0 | 37.5 | 62.5 | 88.9

45. Secondary Outcome: Time to Achieve an F-VASI50: Number of Days From the Date of the First Application in the Double-Blind Period to the Date of the First Evaluation at Which the Participant Met the F-VASI50 Score
Description: as for outcome 14
Time Frame: up to 52 weeks
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved an F-VASI50. | 197.0 [127.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved an F-VASI50. | 339.0 [195.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved an F-VASI50. | 172.0 [127.0 to 323.0] | 170.0 [127.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved an F-VASI50.

46. Secondary Outcome: Time to Achieve a T-VASI50: Number of Days From the Date of the First Application in the Double-Blind Period to the Date of the First Evaluation at Which the Participant Met the T-VASI50 Score
Description: A T-VASI50 responder achieved at least 50% improvement from Baseline in T-VASI. T-VASI was measured by the percentage of vitiligo involvement from all body regions (percentage of BSA; assessed by the Investigator) and the degree of depigmentation: 0% (no depigmentation), 10% (only specks of depigmentation), 25% (pigmented area exceeded depigmented area), 50% (depigmented and pigmented area was equal), 75% (depigmented area exceeded pigmented area), 90% (specks of pigment present), 100% (no pigment present). T-VASI was derived by multiplying the vitiligo involvement values by the percentage of affected skin for each body site and summing all values (possible range: 0-100; lower scores indicate increased improvement).
Time Frame: up to 52 weeks
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved a T-VASI50. | NA [204.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants achieved a T-VASI50. | NA [366.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants achieved a T-VASI50. | NA [192.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants achieved a T-VASI50. | 376.0 [276.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved a T-VASI50.

47. Secondary Outcome: Time to Achieve an F-PhGVA of Clear or Almost Clear
Description: The severity of vitiligo was assessed by the physician using the PhGVA, which has a 5-point scale. 0=clear, no signs of vitiligo; 1=almost clear, only specks of depigmentation present; 2=mild disease, pigmented and depigmented areas are equal; 3=moderate disease, more or complete depigmentation (may include < 30% hair whitening); 4=severe disease, complete depigmentation plus > 30% hair whitening. Time to achieve an F-PhGVA response was defined as the number of days from the date of the first application in the Double-Blind Period to the date of the first evaluation at which the participant met the F-PhGVA score.
Time Frame: up to 52 weeks
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved an F-PhGVA of clear or almost clear. | 372.0 [274.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved an F-PhGVA of clear or almost clear. | NA [369.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants achieved an F-PhGVA of clear or almost clear. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved an F-PhGVA of clear or almost clear. | NA [367.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants achieved an F-PhGVA of clear or almost clear.

48. Secondary Outcome: Time to Achieve an T-PhGVA of Clear or Almost Clear
Description: The severity of vitiligo was assessed by the physician using the PhGVA, which has a 5-point scale. 0=clear, no signs of vitiligo; 1=almost clear, only specks of depigmentation present; 2=mild disease, pigmented and depigmented areas are equal; 3=moderate disease, more or complete depigmentation (may include < 30% hair whitening); 4=severe disease, complete depigmentation plus > 30% hair whitening. Time to achieve a T-PhGVA response was defined as the number of days from the date of the first application in the Double-Blind Period to the date of the first evaluation at which the participant met the T-PhGVA score.
Time Frame: up to 52 weeks
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved a T-PhGVA of clear or almost clear. | 372.0 [274.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved a T-PhGVA of clear or almost clear. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved a T-PhGVA of clear or almost clear. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved a T-PhGVA of clear or almost clear. | NA [369.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants achieved a T-PhGVA of clear or almost clear.

49. Secondary Outcome: Time to Achieve a PaGIC-V of Very Much Improved or Much Improved
Description: The PaGIC-V is an assessment of improvement by the participant. It is a 7-point scale comparing the vitiligo areas at Baseline with the participant's treated areas of vitiligo at the study visit. The participant answered the following: "Since the start of the treatment you've received in this study, your vitiligo in areas treated with the study drug is: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; and 7, very much worse. Time to achieve a PaGIC-V response was defined as the number of days from the date of the first application in the Double-Blind Period to the date of the first evaluation at which the participant met the PaGIC-V score.
Time Frame: up to 52 weeks
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% QD | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
Number analyzed (Participants) | 32 | 31 | 31 | 30 | 33
days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants achieved a PaGIC-V of very much improved or much improved. | NA [274.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants achieved a PaGIC-V of very much improved or much improved. | NA [290.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants achieved a PaGIC-V of very much improved or much improved. | 282.0 [169.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved a PaGIC-V of very much improved or much improved. | 281.0 [178.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants achieved a PaGIC-V of very much improved or much improved.

ADVERSE EVENTS:
Time Frame: Up to 180 weeks (156-week treatment period plus 6-month follow-up period)
Description: 157 participants received 1 of 4 doses of ruxolitinib cream or vehicle during the 24-week, DB period. After the DB period, 11 stayed on 0.15% QD and 42 were re-randomized to 1 of 3 higher groups. All others remained on the same treatment regimen through Week 52. 47 randomized to the 1.5% BID arm during Week 52 stayed during the OL period and 83 from the 3 lower dose arms (0.15% QD, 0.5% QD, and 1.5% QD) crossed over to the 1.5% BID arm during the OL period, totaling 130 at risk at data cut-off.
Groups:
- Ruxolitinib Cream 0.15% Once Daily (QD): All participants who received at least one dose of ruxolitinib cream 0.15% QD (in the 52-week combined vehicle-controlled and continued double-blind periods).
- Ruxolitinib Cream 0.5% QD: All participants who received at least one dose of ruxolitinib cream 0.5% QD. Treatment was received by participants for 52 weeks in the combined vehicle-controlled and continued double-blind periods, and by those participants who were randomized to the vehicle group or were randomized to ruxolitinib cream 0.15% QD and did not achieve 25% improvement in F-VASI score at Week 24 and crossed over to 0.5% QD for 28 weeks (Week 24 to Week 52 [continued double-blind treatment period]).
- Ruxolitinib Cream 1.5% QD: All participants who received at least one dose of ruxolitinib cream 1.5% QD. Treatment was received by participants for 52 weeks in the combined vehicle-controlled and continued double-blind periods, and by those participants who were randomized to the vehicle group or were randomized to ruxolitinib cream 0.15% QD and did not achieve 25% improvement in F-VASI score at Week 24 and crossed over to 1.5% QD for 28 weeks (Week 24 to Week 52 [continued double-blind treatment period]).
- Ruxolitinib Cream 1.5% BID: All participants who received at least one dose of ruxolitinib cream 1.5% BID. Treatment was received by (1) participants randomized to ruxolitinib cream 1.5% BID through Week 156, (2) participants who were randomized to the vehicle group or were randomized to ruxolitinib cream 0.15% QD and did not achieve 25% improvement in F-VASI score at Week 24 and crossed over to 1.5% BID for 28 weeks (Week 24 to Week 52 [continued double-blind treatment period]), and (3) participants who were (a) randomized to the vehicle group, (b) to ruxolitinib cream 0.15% QD and achieved 25% improvement in F-VASI score at Week 24, (c) to ruxolitinib cream 0.5% QD, and (d) to ruxolitinib cream 1.5% QD who crossed over to 1.5% BID during the open-label extension period.
Arm/Group | Vehicle Twice Daily (BID) | Ruxolitinib Cream 0.15% Once Daily (QD) | Ruxolitinib Cream 0.5% QD | Ruxolitinib Cream 1.5% QD | Ruxolitinib Cream 1.5% BID
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/45 | 0/44 | 0/130
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 2/45 | 1/44 | 4/130
Other Adverse Events (participants affected / at risk) | 14/32 | 19/31 | 23/45 | 20/44 | 45/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Twice Daily (BID) (N=32) | Ruxolitinib Cream 0.15% Once Daily (QD) (N=31) | Ruxolitinib Cream 0.5% QD (N=45) | Ruxolitinib Cream 1.5% QD (N=44) | Ruxolitinib Cream 1.5% BID (N=130)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Twice Daily (BID) (N=32) | Ruxolitinib Cream 0.15% Once Daily (QD) (N=31) | Ruxolitinib Cream 0.5% QD (N=45) | Ruxolitinib Cream 1.5% QD (N=44) | Ruxolitinib Cream 1.5% BID (N=130)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (7) | 4 (4) | 5 (12) | 4 (5) | 12 (14)
Application site erythema (General disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Application site exfoliation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Application site pruritus (General disorders) | 3 (3) | 6 (8) | 3 (3) | 3 (4) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 6 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (5) | 5 (6) | 5 (6) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 4 (5)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (3) | 5 (5) | 5 (8) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 9 (11)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (2) | 1 (1) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 5 (5) | 1 (3) | 8 (12)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03099304/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT03099304/SAP_001.pdf